CLINICAL TRIAL: NCT06310434
Title: Analysis of COMPASsion and Humanisation of Adolescents Facing the End-of-life Processes: a Mixed-method Participatory Project
Brief Title: Analysis of COMPASsion and Humanisation of Adolescents Facing the End-of-life Processes.
Acronym: COMPAS
Status: Enrolling by invitation | Type: Observational
Sponsor: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Eva Abad-Corpa, RN, PhD, Head of Advanced Nursing Care Group., Instituto de Salud Carlos III
Other Study IDs: PI23/00409
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Compassion; Death Anxiety; Adolescent Behavior
Keywords: Compassion; Death Anxiety; Multicenter Study; Adolescent; Qualitative Research
MeSH Terms: conditions — Necrophobia; Adolescent Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University adolescents: Adolescents attending a public university that belongs to the same "health area" with similar population characteristics in each province. The inclusion criteria will be students enrolled in different undergraduate studies in a public University (18-23 years old), who don´t need curricular adaptation. We will exclude health science studies because we suppose that they are students who may have worked more on compassionate awareness.
  Interventions: Other: questionnaire; Other: Discussion group; Other: Reflective diary
- High school adolescents: The inclusion criteria will be students enrolled in public secondary schools (12-17 years old), that belong to the same "health area". We also include families and teachers because we understand that their knowledge of the context can support the interventions of change proposals and are consistent with the participatory nature of the project. The inclusion criteria for families are parents, mothers, or legal tutors of minors with communication skills to participate in a group. Finally, all the teachers in every center will be invited to participate in the study.
  Interventions: Other: questionnaire; Other: Discussion group; Other: Reflective diary

INTERVENTIONS:
Other: questionnaire — COOL Scale and DAS
Other: Discussion group — Through discussion groups with students in secondary schools and university separately, a compassionate plan will be designed
  Other Names: PAR
Other: Reflective diary — Students can modify the interventions adapting them to their requirements to get the compassion needed for those in need.

SUMMARY:
The investigators want to work on compassion, understood as the recognition of the suffering of others that motivates us to try to alleviate it. The goal of this Multicenter project, with a mixed sequential transformative methodology, is to analyze the impact of a participatory process of awareness and reflection on compassion, in the face of end-of-life processes, in adolescents aged 12-23 years in 6 Spanish provinces, and to understand how the participatory process can transform and improve their compassion.

As the adolescents must be the protagonists of change, the study will be conducted with students enrolled in one public secondary school and in one degree in a public University, that belongs to the same "health area" in each province. The investigators also include families' and teachers' knowledge of the context because it can support the interventions of change proposals.

Compassion will be assessed using the Compassion for the Lives of Others Scale (COOLS), comprising 26 items. Similarly, adolescents' attitudes toward death are another important concept and will be explored through the Death Anxiety Scale (DAS), which has 15 questions. Both scales will be distributed to the adolescents, requesting their permission anonymously.

After the survey, a second phase will start with a Participatory Action Research (PAR) with different activities. The objective is to generate awareness of the need to improve it, allowing the participants to design the interventions, based on evidence-based proposals (cinema forum, colloquiums with testimonies of volunteers accompanying palliative patients, organization of Death Cafe, artistic and literary activities, generation of grief groups, etc.).

At the end of the project, the investigators will evaluate the adolescent compassion level and create discussion groups again to understand the impact of the interventions.

With this project, the investigators will empower new generations of people to encourage, facilitate, support, and celebrate mutual care and family and community development in end-of-life processes. The translation and implications of the results for clinical practice will contribute to reducing inequalities in health research in a vulnerable group of special interest, especially when treatments can do nothing for their survival but with interventions such as those in this study, the investigators can ensure quality and dignity of life as long as there is life.

DETAILED DESCRIPTION:
A multicenter project is proposed and designed as a mixed methods transformative sequential study in two phases:

PHASE 1, Diagnosis of the situation of compassion, through a descriptive observational study that will provide valuable information about understanding compassionate awareness in adolescents and will be useful for rigorously evaluating changes post-intervention in specific groups.

To analyze the level of compassion of adolescents in every province, the investigators include all the public secondary schools and a public university that belong to the same "health area" with similar population characteristics in each province. In the 6 participating Universities there are 340 degrees and a total of 92103 students enrolled. In the 6 Health Areas of the study provinces, there are 61 high schools and the population of adolescents enrolled in school is 36486. Thus, a random sample of 1852 individuals is enough to estimate, with 95% confidence and a precision of +/- 0.10 units, the population means values that are expected to have a standard deviation of about 1.56 units.

A series of sociodemographic and educational variables will be collected from all participants to describe their characteristics, such as age, gender, level of studies, school, educational context, previous experience with dying people, volunteer activities, or other personal experience in palliative care (PC). Compassion will be assessed using the COOLS and adolescents' attitudes toward death, which will be explored through the DAS. The evaluation scales will be distributed to the adolescents, requesting their permission to distribute the questionnaires anonymously through the different specific communication channels that each educational center (secondary school and university) uses to keep up communication with the students. The responses will be recorded online in the Research Electronic Data Capture (REDCap), an electronic data capture software.

The investigators will elaborate a descriptive summary document on the level of adolescent compassion in all provinces taking into account variables such as educational context, context compassion resources, age, and gender. The investigators will analyze the differential characteristics of sex in compassion from a gender perspective. In general, the investigators will make descriptive statistics according to the nature of the variables with 95% confidence intervals.

PHASE 2, related to the compassion transformation process. To understand how the process of sensitization and participatory reflection is capable of transforming compassion, the investigators design a PAR study based on the proposal of Stephen Kemmis and Robin McTaggart who suggest a PAR that focuses on the collective change that is produced from the individual reflections of the participants in a social context. The research process will be participatory and cooperative to propose and promote effective changes from the participants and their context. The project is designed in a sequence of cycles to design interventions, implementation, and evaluation.

Before the activities, a literature review will be done by the investigators to identify effective interventions to improve compassionate awareness in adolescents used by other researchers. Next, the investigators will design a plan of compassionate good practices in a participatory manner, through discussion groups with students in secondary schools and universities separately. In secondary school, the investigators also will do groups with families and teachers, separately, because they can contribute to adapting these good practices to students' context. In addition, the investigators will propose to the students that they carry out a reflective diary. The objective is to generate awareness of the need to improve it, allowing the participants to design the interventions, based on evidence-based proposals. The participants can modify, adapt, and suggest new interventions participants believe can work out in each center. In the research team, there are professional experts in knowledge transfer and in the adolescent population, therefore, the professional experts will advise on how to present the information to each group, adapting the local language, format, and cultural elements. The research team will also facilitate the mobilization of resources that allow the implementation of the interventions, and when the interventions are implemented, the adolescents' satisfaction will be evaluated with structured surveys.

At the end of the project, the investigators will evaluate the adolescent compassion level, replaying the same process as the beginning of the project (phase 1). Afterward, the investigators will do discussion groups again, to understand better the impact of the interventions on their compassion perception.

Data analysis would be adjusted to PRISMA (Preferred Reporting Items for Systematic Reviews and Meta-Analyses) indications when the literature review is being carried out. Then, discussion groups will be recorded and transcribed, and will do a critical analysis of the discourse. Inductive and deductive strategies will be employed. In the inductive phase, the different levels of units of meaning are identified in an exhaustive and triangulated manner: codes, subcategories, and categories. Each transcribed document will be read and analyzed independently by two researchers. In the deductive phase, the data will be analyzed from the data obtained from the literature review and theoretical framework.

The data were triangulated by two members of the research team and shared. The investigators will work responding to reliability and authenticity criteria suggested by Lincoln and Guba: credibility, transferability, dependency, and confirmability. In addition, the rigor criteria established in COREQ-32 (Consolidated Criteria for Reporting Qualitative Research) were also followed in the design of Phase 2 with qualitative methodology.

The investigators will elaborate a survey ad-hoc, with quantitative and qualitative items, to know participants' satisfaction with the intervention, organization, and their opinions. The qualitative results from the ad-hoc evaluation will be analyzed with a content analysis to assess the relevance, suitability, and impact of each intervention. To understand the changes that the project has caused them, the investigators will do a critical analysis of the discourse of the discussion groups in the evaluation phase.

Before starting the fieldwork, approval will be obtained from the research ethics committee of each province. All participants who wish to be part of the project will voluntarily sign the informed consent. Appropriate anonymization and privacy-preserving methods are employed to ensure the privacy of users when their personally identifiable information is stored, processed, and shared. Special attention and strict legal compliance will be paid to underage adolescent participation. As established by Organic Law 1/1996 -on the Legal Protection of Minors - modified by Law 26/2015 and Law 45/2015 (Spanish laws), the investigators who have any interaction with the minors under study accredit that they have not committed crimes of a sexual nature through a certificate issued by the Spanish Ministry for Justice. The present study will be developed by the Declaration of Helsinki and the Good Clinical Practice Guidelines. Following the protocol and legal requirements specified by Law, 14/2007 on Biomedical Research and the precepts contained in the European Union (EU) Chart of Fundamental Rights (2000/C 364/01) and the EU Regulation 2016/679 of the European Parliament will be complied with. Participants may exercise all their rights under the Statutory Law Protection of Personal Data and Guaranteeing Digital Rights 3/2018 and Data Protection Regulation 2016/679 (Spanish Laws).

Identification of critical points and contingency plan: The population-based survey study has the limitations of observational studies. The fact that members of the educational community recruit and encourage adolescents to participate, minimizes the loss of follow-up. Limitations of qualitative research relate to participation and data collection, therefore, more time may be needed to overcome initial distrust and reluctance to join the research. Taking into account these limitations, the timetable defined has taken into account the characteristics of the population by proposing sufficient time for the PAR process. As with all multicenter projects that focus on complex health and social care interventions, there are potential risks and barriers. The investigators include our contingency plans:

1. Risk of not having consistency of approach between regional institutions (severity: medium risk 20%): To risk mitigation the investigators propose early warning systems with frequent monitoring of data collection processes between partners and feedback on progress is arranged by developing a robust communication system early on that will proactively identify and solve problems.
2. Delays to empirical work (medium risk 20%): The project coordinator is well experienced in guiding these kinds of projects. Moreover, participants are chosen based on their experience in dealing with research in this area and their existing close connections to the site.
3. Risk of not recruiting the minimum participants (medium risk 15%): The commitment made by the participants is for a relatively long period, as PAR is a reflective process that requires at least two full cycles per group. Critical points will be established for scheduling progressive recruitment; therefore, in case some point is not reached, additional units will be recruited within the institutions.
4. High drop-out rate (non-valid results due to lack of a representative number of participants) (medium risk 20%): Critical points will be established taking in that conversation about death is often associated with fear, anxiety, avoidance, and misunderstandings in adolescents. Many adults feel that these discussions are inappropriate and confusing for young people. Before working with teenagers, the investigators will explain the project and get their parents' consent. On the other hand, potential institutions that could be influenced first by project results will be analyzed from the first stages of the project and could be potential collaborators.
5. Shortage of resources (medium risk 20%): Consortium agreement between all researchers binds them concerning the availability of resources. Early warning systems of monthly time reporting and 6-monthly financial reporting allow to detect problems timely and take action.
6. Dissemination activity is ineffective at increasing the visibility of the Project (low risk 5%): A dissemination strategy is developed early in the project to identify the correct audience and devise strategies to reach them.
7. Insufficient interaction with targeted communities (low risk 5%): Increase the presence of representatives of the target groups in all stages of the project, including the exploitation activities. Step up the communication in case of not satisfying the target communities, intensifying the communication and adapting it even more to their specific needs.

These plans are based on tried and tested strategies, from previous projects and international implementation papers, and the investigators are confident of their robustness. In addition, the investigators will have an Internal Executive Quality Assurance group within the team whose responsibilities will include four-month assessments of project delivery, which will enable the investigators to pre-empt and tackle problems before they arise.

ELIGIBILITY:
Inclusion Criteria:

* University and high schools that belong to the same "Health Area"
* Students enrolled in public secondary schools (12-17 years old) and in different undergraduate studies in a public University (18-23 years old) during the development of the project
* Parents, mothers, or legal tutors of minors with communication skills to participate in a group

Exclusion Criteria:

* Students who need curricular adaptation
* Health science studies at the University

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The project will be conducted in six "Health Areas" in 6 Spanish provinces: Baleares, Barcelona, Madrid, Murcia, Huelva, and Málaga. In each province, we will include all the public secondary schools and a public university that belong to the same "Health Area" with similar population characteristics in each province. In the 6 participating Universities there are 340 degrees and a total of 92103 students enrolled. In the 6 "Health Areas" of the study provinces, there are 61 high schools and the enrolled adolescents in school are 36486 students.
Sampling Method: Probability Sample
Enrollment: 1852 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Describe and improve the level of compassion of high school and university students. | first 8 weeks and the last 8 weeks of the academy year
  Compassion is understood as the recognition of the suffering of others that motivates us to try to alleviate it. Compassion will be assessed using the "Compassion for the Lives of Others Scale" (COOL Scale), which comprises 26 items, of which 13 correspond to the empathy dimension and the remaining 13 to the relief of suffering dimension, presented on a 7-point Likert scale format, graded according to agreement with the statement (from 1 = strongly disagree to 7 = strongly agree). The scale provides an overall score for the degree of compassion towards others as well as a score for each subscale (empathy and relief of suffering).
Describe and improve the attitude towards death of high school and university students. | first 8 weeks and the last 8 weeks of the academy year
  The Death Anxiety Scale (DAS) assesses "fear of death, fear of illness, preoccupation with time, preoccupation with death", it comprises 15 self-administered dichotomous (true or false) response items. Items 1, 4, 8, 9, 10, 11, 12, 13, and 14 are scored 1 point if the answer is true and 0 points if it is false; conversely, the other six items, 2, 3, 5, 6, 7, and 15, are scored 1 point if the answer is false. The range of total scores for Death Anxiety was between 0 and 15, with higher scores indicating higher Death Anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Abad-Corpa, PhD, Principal Investigator — Instituto Murciano de Investigación Biosanitaria
Locations (1):
- Instituto Murciano de Investigación Biosanitaria, Murcia, MU, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data will be used exclusively for the purposes of the COMPAS study. Data will be shared with collaborators under confidentiality agreements. In scientific publications, data will be presented in aggregate form without any possibility of participant identification.
  Consideration will be given to sharing anonymized quantitative data in an open-access repository and on platforms such as Zenodo and Open Research Europe, subject to approval by the ethics committee and with the consent of participants.
  Publication of research results in open-access scientific journals. Presentation of results at conferences and seminars.

REFERENCES:
- [Background] Abel J. Compassionate communities and end-of-life care. Clin Med (Lond). 2018 Feb;18(1):6-8. doi: 10.7861/clinmedicine.18-1-6. PMID 29436431
- [Background] Kellehear, A. Lowton, Karen. Compassionate Cities. Public Health and End of Life Care. Sociology of health & illness Volume: 30 Issue 1 (2008) ISSN: 0141-9889
- [Background] Abel J, Bowra J, Walter T, Howarth G. Compassionate community networks: supporting home dying. BMJ Support Palliat Care. 2011 Sep;1(2):129-33. doi: 10.1136/bmjspcare-2011-000068. PMID 24653223
- [Background] Vanderstichelen S. Palliative care volunteering: Pressing challenges in research. Palliat Med. 2022 Apr;36(4):564-566. doi: 10.1177/02692163221089483. Epub 2022 Mar 31. No abstract available. PMID 35360995
- [Background] Soderhamn U, Flateland S, Fensli M, Skaar R. To be a trained and supported volunteer in palliative care - a phenomenological study. BMC Palliat Care. 2017 Mar 14;16(1):18. doi: 10.1186/s12904-017-0193-0. PMID 28288598
- [Background] Chambers E, Gardiner C, Thompson J, Seymour J. Patient and carer involvement in palliative care research: An integrative qualitative evidence synthesis review. Palliat Med. 2019 Sep;33(8):969-984. doi: 10.1177/0269216319858247. Epub 2019 Jun 28. PMID 31250702
- [Background] Hasson N, Urtaran-Laresgoiti M, Nuno-Solinis R, Moreno I, Espiau G, Grajales M, Fonseca J. Community Based Participatory Research For The Development of a Compassionate Community: The Case of Getxo Zurekin. Int J Integr Care. 2022 Jan 17;22(1):2. doi: 10.5334/ijic.5707. eCollection 2022 Jan-Mar. PMID 35087351
- [Background] Librada-Flores S, Nabal-Vicuna M, Forero-Vega D, Munoz-Mayorga I, Guerra-Martin MD. Implementation Models of Compassionate Communities and Compassionate Cities at the End of Life: A Systematic Review. Int J Environ Res Public Health. 2020 Aug 28;17(17):6271. doi: 10.3390/ijerph17176271. PMID 32872244
- [Background] Dumont K, Marcoux I, Warren E, Alem F, Alvar B, Ballu G, Bostock A, Cohen SR, Daneault S, Dube V, Houle J, Minyaoui A, Rouly G, Weil D, Kellehear A, Boivin A. How compassionate communities are implemented and evaluated in practice: a scoping review. BMC Palliat Care. 2022 Jul 20;21(1):131. doi: 10.1186/s12904-022-01021-3. PMID 35854292
- [Background] Bakelants H, Vanderstichelen S, Chambaere K, Van Droogenbroeck F, De Donder L, Deliens L, Dury S, Cohen J. Researching Compassionate Communities: Identifying theoretical frameworks to evaluate the complex processes behind public health palliative care initiatives. Palliat Med. 2023 Feb;37(2):291-301. doi: 10.1177/02692163221146589. Epub 2022 Dec 28. PMID 36576313
- [Background] Zarco Colón, J., Ramasco Gutiérrez, M., Pedraz Marcos, A., & Palmar Santos, A. M. (2019). Investigación cualitativa en salud (Vol. 58). CIS.
- [Background] Ivankova, N. (2017). Applying mixed methods in community-based participatory action research: a framework for engaging stakeholders with research as a means for promoting patient-centredness. Journal of Research in Nursing, 22 (4), 282-294.
- [Background] Ivankova, N., & Wingo, N. (2018). Applying mixed methods in actions research: methodological potentials and advantages. American Behavioral Scientist, 62(7), 978-997.
- [Background] Farquhar MC, Ewing G, Booth S. Using mixed methods to develop and evaluate complex interventions in palliative care research. Palliat Med. 2011 Dec;25(8):748-57. doi: 10.1177/0269216311417919. Epub 2011 Aug 1. PMID 21807749
- [Background] Fabregues S, Hong QN, Escalante-Barrios EL, Guetterman TC, Meneses J, Fetters MD. A Methodological Review of Mixed Methods Research in Palliative and End-of-Life Care (2014-2019). Int J Environ Res Public Health. 2020 May 29;17(11):3853. doi: 10.3390/ijerph17113853. PMID 32485830
- [Background] Tashakkori A, Teddlie C. (2012). Utilizing mixed-methods in psychological research. Weiner, I, Schinka JA, Velicer WF. Handbook of Psychology, Research Methods in Psychology. (N.º 2 edición. (19 octubre 2012). Wiley.
- [Background] Kemmis S, McTaggart R, Nixon R. The action research planner: Doing critical participatory action research. The Action Research Planner: Doing Critical Participatory Action Research. 2014. 1-200 p.
- [Background] Chang, Fresco, & Green. The Development and Validation of the Compassion of Others' Lives Scale (The COOL Scale). International Journal of Humanities and Social Science. 2014; 4 (5): 33-42.
- [Background] Klos, M. C., & Lemos, V. N. (2018). Adaptación y validación de un instrumento para evaluar el constructo compasión. Revista Evaluar, 18(2), 31-44. Recuperado de https://revistas.unc.edu.ar/index.php/revaluar
- [Background] Tomas-Sabado J, Gomez-Benito J. Psychometric properties of the Spanish form of Templer's Death Anxiety Scale. Psychol Rep. 2002 Dec;91(3 Pt 2):1116-20. doi: 10.2466/pr0.2002.91.3f.1116. PMID 12585522
- [Background] Armas-Arraez MM, Alegre-De la Rosa O, Gutierrez-Barroso J. International Journal of Developmental and Educational Psychology. INFAD Revista de Psicología, Nº1 - Volumen 2, 2021. pp:83-96
- [Background] Abad Corpa E, Delgado Hito P, Cabrero García J. La investigación-acción-participativa: Una forma de investigar en la práctica enfermera. Investig y Educ en Enfermería. 2010;28(3):464-74.
- See also: World Health Organization (WHO) palliative care, facts and figures — https://www.who.int/es/news-room/fact-sheets/detail/palliative-care